CLINICAL TRIAL: NCT05363306
Title: Influence of the Apico-coronal Position of Tissue-level Implants on Marginal Bone Stability
Brief Title: Apico-coronal Position of Tissue-level Implants Bone Stability
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Sponsor
Other Study IDs: TLMBS
Record Dates: First submitted 2022-04-07; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Bone Atrophy, Alveolar
Keywords: osseointegrated implant; early marginal bone loss;
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- thin crestal mucosa: Based upon vertical mucosa thickness measured at implant placement, implants were placed: 2mm below the crestal bone in presence of thin mucosa (< 2.5mm)
  Interventions: Procedure: implant insertion
- medium crestal mucosa: Based upon vertical mucosa thickness measured at implant placement, implants were placed: 2) 1mm below the crestal bone in presence of medium mucosa (2.5-3.5mm);
  Interventions: Procedure: implant insertion
- thick crestal mucosa: Based upon vertical mucosa thickness measured at implant placement, implants were placed: 1) at crestal level in presence of thick mucosa (> 3.5 mm);
  Interventions: Procedure: implant insertion

INTERVENTIONS:
Procedure: implant insertion — 4% articaine solution, a mid-crestal incision along the center of the edentulous bone ridge was performed. A full-thickness flap was elevated. The sites were prepared to permit insertion of transmucosal, external hex, implants (I-smart, I-RES, Lugano, Switzerland) at three different crestal levels, based upon vertical mucosa thickness measured at implant placement.
  Owing to width crest, all implants were 3.75 mm in diameter and operators selected appropriate implant lengths (8, 10 mm) according to available bone crest height. All implants were not submerged and flaps were sutured around the transmucosal component.

SUMMARY:
early marginal bone loss around dental implants may hamper long term prognosis of implant-prosthetic rehabilitation. this study aimed to study the correlation of pico-coronal position of dental implant (from supracrestal, crystal to undergone level) measuring early marginal bone loss through periapical x-ray at surgical time and subsequent follow-ups.

DETAILED DESCRIPTION:
Early marginal bone loss (EMBL) is a non-infective remodeling process of peri-implant crestal bone occurring within the first year after implant insertion. EMBL has a multifactorial etiology, being influenced by various surgical and prosthetic factors, including insufficient crestal width, surgical trauma, biological width formation, microbial colonization of implant-abutment micro-gap, horizontal implant-abutment mismatch ("the platform-switching concept"), the number of abutment connection/disconnections, prosthetic abutment height, design and mechanical stability of implant-abutment connection and adaptive response to occlusal loading.

Biological width formation is the main factor influencing peri-implant marginal bone adaptive processes prior to prosthesis delivery. When an implant gets exposed to the oral cavity, soft tissues establish a cuff-like barrier sealing the trans-epithelial component of the fixture.

Differently from equicrestal and subcrestal implants, which present a microgap between implant and abutment at the marginal bone level, tissue-level implants have no gap at this region.

The present multicenter prospective study aims to evaluate if EMBL occurring around tissue-level dental implants before prosthesis delivery may be reduced by adapting apico-coronal positioning in relation to supracrestal tissue thickness.

All patients are treated according to one-stage implant. Sutures are removed 12-14 days after surgery. No removable prostheses are utilized during the healing period.

Final impressions were taken five months after the implant placement. After functional and aesthetic try-in, a single-unit screw-retained metal ceramic crown is delivered. The fixation screw was torqued to 30Ncm following manufacturer's guidelines. Screw access is then closed using light-cured composite resin.

Radiographic measurements. Digital radiographs, customized for each patient with a bite jig, are taken using a long-cone paralleling technique with a film holder at the time of implant placement (baseline, T0), 3 months after implant placement (T1), and 5 months after implant placement, immediately before impression taking (T2). All radiographs are performed using the same x-ray generator technology, set with the same parameters (60 kV, 7 mA).

Two different types of bone changes are calculated, as suggested elsewhere.

1. Early marginal bone loss (EMBL) is calculated.
2. Bone Loss Exposing Implant Surface (BLEIS) is calculated as the difference between the EMBL measurement and the 3 mm length of the transmucosal, machined portion of the implant.

Radiographs demonstrating any deformation, darkness and/or other problem are immediately repeated. All measurements are made by a single calibrated examiner, blind to mucosal thickness, using a 30-inch led-backlit color diagnostic display with Kodak Digital Imaging Software. Each measurement is repeated three times at three different time points as proposed by Gomez-Roman and Launer. Intra-examiner and inter-examiner concordances are 96.1% and 90.4%, respectively, for linear measurements within ±0.1mm.

ELIGIBILITY:
Inclusion Criteria:

* Patients were partially edentulous and required placement of at least one single delayed implant in pristine bone in the posterior mandible
* presence of keratinized mucosa with a minimum bucco-lingual width of 3 mm;
* bone crest with at least 6mm of width and 9 mm of height above the mandibular canal without concomitant or previous bone augmentation procedures;
* presence of the opposing dentition

Exclusion Criteria:

* smokers
* uncontrolled periodontitis
* medication consumption for at least 3 months prior to treatment
* history of head or neck radiation therapy
* pregnancy or lactating at any time during the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were partially edentulous and required placement of at least one single delayed implant in pristine bone in the posterior mandible
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
early marginal bone loss | 5 months after implant placement
  distance from crystal bone to most coronal bone to implant contact

SECONDARY OUTCOMES:
biological complications | during surgery
  any surgical complication

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lombardi, Dr., Principal Investigator — Hesire dental office
Locations (2):
- Italy (2):
  - Hesire, Cassano Allo Ionio, CS
  - Piezosurgery Academy, Parma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lombardi T, Berton F, Salgarello S, Barbalonga E, Rapani A, Piovesana F, Gregorio C, Barbati G, Di Lenarda R, Stacchi C. Factors Influencing Early Marginal Bone Loss around Dental Implants Positioned Subcrestally: A Multicenter Prospective Clinical Study. J Clin Med. 2019 Aug 4;8(8):1168. doi: 10.3390/jcm8081168. PMID 31382675
- [Derived] Spinato S, Bernardello F, Stacchi C, Soardi CM, Messina M, Rapani A, Lombardi T. Marginal Bone Changes Around Tissue-Level Implants After Prosthesis Delivery: A Multicenter Prospective Study. Clin Implant Dent Relat Res. 2025 Jun;27(3):e70071. doi: 10.1111/cid.70071. PMID 40500982